CLINICAL TRIAL: NCT03399578
Title: A Phase I Study to Determine the Safety and Immunogenicity of the Candidate Middle East Respiratory Syndrome Coronavirus (MERS-CoV) Vaccine ChAdOx1 MERS in UK Healthy Adult Volunteers
Brief Title: Safety and Immunogenicity of a Candidate MERS-CoV Vaccine (MERS001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The scientific questions proposed remain relevant, but will now be addressed in a larger phase II immunogenicity trial of the ChAdOx1 MERS vaccine given at 2 doses.
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MERS001
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: MERS (Middle East Respiratory Syndrome)
MeSH Terms: conditions — Coronavirus Infections | interventions — Middle East respiratory syndrome vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): Group 1 volunteers (n= 6) will be administered ChAdOx1 MERS, 5 x 10^9 vp through intramuscular route.
  Interventions: Biological: ChAdOx1 MERS
- Group 2 (Experimental): Group 2 volunteers (n= 9) will be administered ChAdOx1 MERS, 2.5 x 10^10 vp through intramuscular route.
  Interventions: Biological: ChAdOx1 MERS
- Group 3 (Experimental): Group 3 volunteers (n= 9) will be administered ChAdOx1 MERS, 5 x 10^10 vp through intramuscular route.
  Interventions: Biological: ChAdOx1 MERS
- Group 4 (Experimental): Group 4 volunteers (n=6-12) will be administered ChAdOx1 MERS, 2.5 x 10^10 vp at week 0, followed by ChAdOx1 MERS, 2.5 x 10^10 vp at week 26. Both administrations will be given through intramuscular route.
  Interventions: Biological: ChAdOx1 MERS
- Group 5 (Experimental): Group 5 volunteers (n=6-12) will be administered ChAdOx1 MERS, 2.5 x 10^10 vp at week 0, followed by ChAdOx1 MERS, 2.5 x 10^10 vp at week 4. Both administrations will be given through intramuscular route.
  Interventions: Biological: ChAdOx1 MERS

INTERVENTIONS:
Biological: ChAdOx1 MERS — The ChAdOx1 MERS vaccine consists of the replication-deficient simian adenovirus vector ChAdOx1, containing the MERS Spike protein antigen.

SUMMARY:
This is a clinical trial in which healthy volunteers will be administered an experimental MERS vaccine. The vaccine ChAdOx1 MERS will be administered alone both as a single administration and with a homologous prime-booster.

DETAILED DESCRIPTION:
All vaccinations will be administered intramuscularly. In Groups 1-3, each volunteer will receive one vaccination in total. In Groups 4 and 5, each volunteer will receive two vaccinations in total.

There are five different vaccine schedules:

Group 1 (n=6) will receive 5 x 10^9 vp ChAdOx1 MERS .

Group 2 (n=9) will receive 2.5 x 10^10 vp ChAdOx1 MERS.

Group 3 (n=9) will receive 5 x 10^10 vp ChAdOx1 MERS.

Group 4 (n=6-12) will receive 2.5 x 10^10 vp ChAdOx1 MERS at week 0 followed by a boost of 2.5 x 10^10 vp ChAdOx1 MERS at week 26.

Group 5 (n=6-12) will receive 2.5 x 10^10 vp ChAdOx1 MERS at week 0 followed by a boost of 2.5 x 10^10 vp ChAdOx1 MERS at week 4.

The study will assess the safety of the vaccines, and the immune responses to the vaccinations. Immune responses are measured by tests on blood samples.

Healthy adult volunteers will be recruited in Oxford, England.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

1. Healthy adults aged 18 to 50 years
2. Able and willing (in the Investigator's opinion) to comply with all study requirements
3. Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner or access this medical history electronically.
4. For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of screening and vaccination
5. Agreement to refrain from blood donation during the course of the study
6. Provide written informed consent

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
2. Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccine).
3. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
4. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
5. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
6. Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
7. Any history of anaphylaxis in relation to vaccination
8. Pregnancy, lactation or willingness/intention to become pregnant during the study
9. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
10. History of serious psychiatric condition likely to affect participation in the study
11. Bleeding disorder (eg. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
12. Any other serious chronic illness requiring hospital specialist supervision
13. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
14. Suspected or known injecting drug abuse in the 5 years preceding enrolment
15. Seropositive for hepatitis B surface antigen (HBsAg)
16. Seropositive for hepatitis C virus (antibodies to HCV)
17. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
18. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
19. Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate
20. Prior exposure to MERS-CoV (serology will be requested at the discretion of the investigator)
21. History of allergic reaction to Aminoglycoside antibiotics

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited and unsolicited local and systemic adverse events | up to 28 days following vaccination
  The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events. Change from baseline for safety laboratory measures will also be collected. Occurrence of serious adverse events will be collected during the whole study duration

SECONDARY OUTCOMES:
Measures of immunogenicity to the ChAdOx1 MERS vaccine | 12 months
  ELISA to quantify antibodies to MERS Spike protein antigen Ex vivo ELISpot responses to MERS Spike protein antigen

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V Hill, DPhil FRCP, Principal Investigator — Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Folegatti PM, Bittaye M, Flaxman A, Lopez FR, Bellamy D, Kupke A, Mair C, Makinson R, Sheridan J, Rohde C, Halwe S, Jeong Y, Park YS, Kim JO, Song M, Boyd A, Tran N, Silman D, Poulton I, Datoo M, Marshall J, Themistocleous Y, Lawrie A, Roberts R, Berrie E, Becker S, Lambe T, Hill A, Ewer K, Gilbert S. Safety and immunogenicity of a candidate Middle East respiratory syndrome coronavirus viral-vectored vaccine: a dose-escalation, open-label, non-randomised, uncontrolled, phase 1 trial. Lancet Infect Dis. 2020 Jul;20(7):816-826. doi: 10.1016/S1473-3099(20)30160-2. Epub 2020 Apr 21. PMID 32325038